CLINICAL TRIAL: NCT00875771
Title: Phase II Study of Irinotecan, Capecitabine and Bevacizumab in Metastatic Colorectal Cancer Patients
Brief Title: Irinotecan, Capecitabine and Bevacizumab in Metastatic Colorectal Cancer Patients
Acronym: AVAXIRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTD-08-03; EudraCT number:2008-004688-20
Record Dates: First submitted 2009-03-30; First posted 2009-04-03 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer; BEVACIZUMAB; CAPECITABINE; IRINOTECAN
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): * Capecitabine: 1000 mg/m2, bid, oral, days 2-8. Every 2 weeks
  * Irinotecan: 175 mg/m2, iv infusion 90 minutes, day 1, every 2 weeks
  * Bevacizumab: 5 mg/kg day 1, every 2 Weeks
  Interventions: Drug: Capecitabine+Irinotecan+Bevacizumab

INTERVENTIONS:
Drug: Capecitabine+Irinotecan+Bevacizumab — * Capecitabine: 1000 mg/m2, bid, oral, days 2-8. Every 2 weeks
  * Irinotecan: 175 mg/m2, iv infusion 90 minutes, day 1, every 2 weeks
  * Bevacizumab: 5 mg/kg day 1, every 2 Weeks
  Treatment will be given until disease progression or unacceptable toxicity.

SUMMARY:
The purpose of this study is to determine efficacy and safety of the biweekly scheme with Capecitabine and Irinotecan, plus bevacizumab in patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
The purpose of this study is to determine efficacy and safety of the biweekly scheme with Capecitabine and Irinotecan, plus bevacizumab in patients with metastatic colorectal cancer.

* Capecitabine: 1000 mg/m2, bid, oral, days 2-8. Every 2 weeks
* Irinotecan: 175 mg/m2, iv infusion 90 minutes, day 1, every 2 weeks
* Bevacizumab: 5 mg/kg day 1, every 2 Weeks

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old (men and women)
2. ECOG Performance Status ≤ 2.
3. Histologically confirmed colorectal adenocarcinoma, metastatic disease.
4. No surgery option
5. No previous chemotherapy, except adjuvant treatment finished at least 6 months before the study inclusion
6. Have at least one measurable lesion according to the RECIST criteria
7. At least a 3-month life expectancy.
8. Written informed consent given.

Exclusion Criteria:

1. Patients who have previously received systemic treatment (for example, cytostatic chemotherapy or active/passive immunotherapy) for advanced or metastatic disease.
2. Patients previously treated with bevacizumab
3. Prior adjuvant or neoadjuvant treatment for non-metastatic disease (M0) is allowed, as long as it has concluded at least 6 months before beginning the treatment of the study.
4. If adjuvant treatment has previously been administered, the patients cannot have shown progression of the disease during treatment nor during the 6 months following termination thereof.
5. Prior radiotherapy is allowed if it has not been administered in the target lesions selected for this study, unless progression of said lesions in the irradiated field is documented, and as long as treatment has concluded at least 4 weeks before beginning the study.
6. Prior surgical treatment of the disease in stage IV is allowed.
7. Only non evaluable disease (non measurable) as ascitis, pleural effusion, diffuse hepatic, osseous metastasis
8. History of another neoplastic disease during the last five years, with the exception of cured basal cell carcinoma of the skin and cervical carcinoma in situ.
9. History or indications of CNS disease (for example, primary brain tumor, uncontrolled convulsions with standard medical treatment, cerebral metastases of any type or history of ictus) in the physical examination.
10. Medication or peripheral vascular disease, grade II or higher. Furthermore, those patients who have had a myocardial infarction in the year prior to beginning the treatment of the study will be excluded.
11. History of psychiatric disability that the investigator considers clinically significant, which prevents the patient from granting the informed consent or interferes with compliance of taking the oral medication
12. Clinically significant cardiovascular disease (i.e., active), for example, uncontrolled hypertension, unstable angina, congestive heart failure, class II or higher of the New York Heart Association (NYHA), severe cardiac arrhythmia
13. Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome or inability to take oral medication.
14. Patients subjected to organ allografts who require immunosuppressive treatment.
15. Severe, non-cicatrized osseous fractures, wounds or ulcers.
16. Indications of hemorrhagic diathesis or coagulopathy.
17. Severe, uncontrolled intercurrent infections or other severe, uncontrolled concomitant diseases.
18. Moderate or severe renal failure [creatinine clearance lower than 30 ml/min (calculated according to the Cockcroft-Gault Formula)] or serum creatinine > 1.5 x upper limit of normal (ULN).
19. Any of the following laboratory values:

    * Absolute neutrophils count (ANC) ≤ 1.5 x 109/l.
    * Platelet count ≤ 100 x 109/l.
    * Hemoglobin ≤ 9 g/dl.
    * INR > 1.5.
    * Total bilirubin >1.5 ULN.
    * ALS and/or AST > 2.5 x ULN or > 5 x ULN (in case of hepatic metastasis).
    * Alkaline phosphatase > 2.5 x ULN or 5 x ULN (in case of hepatic metastasis), or > 10 x ULN (in case of bone metastasis).
20. History of unexpected serious adverse events to fluoropyrimidine treatments or known dihidropyrimidine dehydrogenase (DPD) deficiency.
21. Patients subjected to major surgical procedure, open biopsy or patients have been significant traumatic injures in 28 days time before the initial study treatment, or patients with a major surgery procedure planning during the study period. Fine needle aspiration biopsy 7 days before the initial study.
22. Use of full dose of oral or parenteral anticoagulants ( at least 10 days before the initial study treatment or thrombolytic agents. Low dose of warfarin is allowed, with an INR ≤ 1.5
23. Subject requiring chronic use of high dose aspirin (> 325 m/day) or non-steroidal anti-inflammatory treatment (those known to inhibit platelet function at doses used to treat chronic inflammatory diseases).
24. Pregnant (serum positive pregnancy test) or lactating women.
25. Received any investigational drug or agent/ procedure, i.e. participation in another treatment trial within 30 days of randomisation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 2009-2012

SECONDARY OUTCOMES:
overall survival (SG) | 2009-2012
Overall Response rate | 2009-2012
Toxicity | 2009-2012
Duration of response | 2009-2012
Quality of life | 2009-2012
Rate of hepatic metastases resection | 2009-2012

CONTACTS AND LOCATIONS:
Overall Officials: Pilar García Alfonso, MD, Study Chair — Hospital Gregorio Marañón. Madrid. Spain; Enrique Aranda, MD; phD, Study Chair — Hospital Reina Sofía. Cordoba. Madrid
Locations (1):
- Spanish Cooperative Group for Gastrointestinal Tumour Therapy, Madrid, Spain

REFERENCES:
- [Derived] Garcia-Alfonso P, Chaves M, Munoz A, Salud A, Garcia-Gonzalez M, Gravalos C, Massuti B, Gonzalez-Flores E, Queralt B, Lopez-Ladron A, Losa F, Gomez MJ, Oltra A, Aranda E; Spanish Cooperative Group for the Treatment of Digestive Tumors (TTD). Capecitabine and irinotecan with bevacizumab 2-weekly for metastatic colorectal cancer: the phase II AVAXIRI study. BMC Cancer. 2015 Apr 29;15:327. doi: 10.1186/s12885-015-1293-y. PMID 25925749
- See also: Related Info — http://www.ttdgroup.org